CLINICAL TRIAL: NCT01484262
Title: Liraglutide or Insulin in Real Life Usage in Patients With Diabetes Mellitus Type 2
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-3962; U1111-1123-5044 (Other: WHO)
Record Dates: First submitted 2011-11-22; First posted 2011-12-02 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Liraglutide
  Interventions: Drug: liraglutide
- Any insulin
  Interventions: Drug: insulin

INTERVENTIONS:
Drug: liraglutide — Patients will be treated according to routine clinical practice at the discretion of the treating physician according to current labelling.
  Groups: Liraglutide
Drug: insulin — Any insulin in any device available on the market may be used by patients as part of routine clinical practice according to current labelling.
  Groups: Any insulin

SUMMARY:
This study is conducted in Europe. The intention of this health service research study is to obtain data from daily routine to evaluate the quality of life and the costs of the disease for patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. (Study-related activities are any procedures related to recording of data according to the protocol)
* Patients willing and able to give signed consent on matching patient data with sick fund data
* Patients diagnosed with type 2 diabetes mellitus, currently treated with oral antidiabetic medication, who need treatment intensification with insulin or liraglutide (Victoza®) due to inadequate blood glucose control
* Patient is a member of the involved sick fund (AOK Plus)

Exclusion Criteria:

* Known or suspected contra-indication to the relevant study product according to current SPC
* Previous participation in this study
* History of type 1 diabetes mellitus
* Previous insulin treatment excluding emergency administration (treatment duration up to a maximum of 3 days)
* Previous treatment with liraglutide
* History of diabetic gastroparesis, diabetic precoma or diabetic ketoacidosis
* Progressive fatal disease
* Any reason in judgement of the treating physician that precludes study participation e.g. lack of compliance, safety concerns, alcohol or drug abuse
* Patients without legal capacity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with type 2 diabetes mellitus, currently treated with oral antidiabetics (OADs), who need treatment intensification with insulin or liraglutide due to inadequate blood glucose control.
Sampling Method: Non-Probability Sample
Enrollment: 1344 (Actual)
Dates: Start 2011-11-14 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2014-10-31 (Actual)

PRIMARY OUTCOMES:
Diabetes-related quality of life assessed by ADDQoL (Audit of Diabetes-Dependent Quality of Life) | At the end of the observational period (52 weeks)

SECONDARY OUTCOMES:
Total cost of patient's diseases | At the end of the observational period (52 weeks)
Total cost of patient education | At the end of the observational period (52 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Mainz, Germany

REFERENCES:
- [Result] Lundershausen R, Muller S, Hashim M, Kienhofer J, Kipper S, Wilke T. Quality of Life, Glycemic Control, Safety and Tolerability Associated with Liraglutide or Insulin Initiation in Patients with Type 2 Diabetes in Germany: Results from the Prospective, Non-interventional LIBERTY Study. Exp Clin Endocrinol Diabetes. 2020 Mar;128(3):170-181. doi: 10.1055/a-0636-3961. Epub 2018 Aug 29. PMID 30157532
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com